CLINICAL TRIAL: NCT01811134
Title: Multicenter Randomized Study for Medico-economic Evaluation of Embolization With Flow Diverter Stent in the Endovascular Treatment of Unruptured Saccular Wide-necked Intracranial Aneurysms
Brief Title: Flow Diverter Stent for Endovascular Treatment of Unruptured Saccular Wide-necked Intracranial Aneurysms
Acronym: EVIDENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011.689; 2011-A01079-32 (Other: IDRCB)
Record Dates: First submitted 2012-11-20; First posted 2013-03-14 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Intracranial Aneurysm
Keywords: endovascular procedure; flow diverter stent
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PIPELINE flow diverter stent (Experimental): flow diverter stent
  Interventions: Device: PIPELINE flow diverter stent; Device: Coils, with or without expendable stent
- Coils, with or without expendable stent (Active Comparator): Coils
  Interventions: Device: PIPELINE flow diverter stent; Device: Coils, with or without expendable stent

INTERVENTIONS:
Device: PIPELINE flow diverter stent — endovascular procedure using the medical device PIPELINE
Device: Coils, with or without expendable stent — endovascular embolization procedure using microspires, with the possibility of using a balloon temporary and / or implantation of a stent complementary intracranial before implementation of microspires

SUMMARY:
Unruptured saccular intracranial aneurysms larger than 7 mm can be treated with endovascular occlusion using detachable coils, with or without expendable stent assistance. A new endovascular technique has recently been developed, using flow diverter stents without associated coils. Clinical results already published are encouraging but have to be confirmed. Furthermore, these medical devices are expensive in comparison to the coiling strategy. The purpose of this study is to compare the clinical efficacy, safety, and cost-effectiveness of endovascular coiling and endovascular flow diversion for unrupted saccular intracranial aneurysms.

DETAILED DESCRIPTION:
Main Outcome Measure: Percentage of patients with an aneurysm with complete occlusion, defined as the absence of visible blood flow to the consideration of angiography performed 12 months post-endovascular intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age ≥ 18 years old
* Unruptured saccular intracranial aneurysm diagnosed by angiography or CT angiography or MR angiography, located in the intra-dural area, with a neck diameter between 4 and 10 mm, with a sac diameter between 7 mm and 20 mm, with a ratio "dome/nek" greater than 1, and with a diameter of the parent artery between 2 and 5 mm.
* No prior treatment of the aneurysm
* Agreement for participating in the study and informed consent signed by the patient
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patient's age < 18 years old
* Adult patient protected by law
* Contraindications to the endovascular procedure
* Contraindications to antiplatelet or anticoagulant treatment
* Prior treatment of the aneurysm
* Presence of an arteriovenous malformation
* Extradural location of the aneurysm
* Fusiform aneurysm
* Active bacterial infection (clinical signs)
* Intracranial hemorrhage from aneurysm in the previous month
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with complete occlusion of the treated aneurysm, defined as the absence of visible blood flow on angiography performed 12 months after endovascular procedure. | 12 months

SECONDARY OUTCOMES:
Occurrence of a death during or after endovascular procedure | hospitalization for the endovascular procedure, up to 7 days
Occurrence of a death whatever the cause | 24 months
Occurrence of a death due to aneurysm rupture | 24 months
Occurrence of an intracranial hemorrhagic from rupture of the aneurysm | 24 months
Occurrence of an ischemic stroke due to thrombosis | 24 months
Occurrence of a non-cerebral bleeding | 24 months
Rate of patients with neurological deficits by mass effect | hospitalization for the endovascular procedure, an expected average of 1 hour; 3 months, 6 months and 12 months post-intervention
Retreatment of the aneurysm | 24 months
Rate of technical complications | Endovascular procedure an expected average of 1 hour
Rate of thromboembolic complications, intraoperative ruptures, complications at the puncture site, or others | Endovascular procedure an expected average of 1 hour
Rate of correct placement of flow diverter stents, according to the investigator | Endovascular procedure an expected average of 1 hour
mean duration of irradiation related to angiography | Endovascular procedure an expected average of 1 hour
Rate of patients for each class of occlusion | Endovascular procedure , an expected average of 1 hour and 12 months
  The classes of occlusion are defined as : complete occlusion, residual neck, residual aneurysm, for the group treated with coiling procedure; grades 0 to 4 according to the scale of Kamran, for the group treated with flow diversion
Modified Rankin score | Inclusion, 3 months and 12 months
National Institute of Health Stroke Score (NIHSS) | Inclusion, 3 months and 12 months
Evolution of the Barthel index | : Inclusion and 12 months
Incremental cost-effectiveness ratio | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francis TURJMAN, PH, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, BRON, France

REFERENCES:
- [Result] Turjman F, Levrier O, Combaz X, Bonafe A, Biondi A, Desal H, Bracard S, Mounayer C, Riva R, Chapuis F, Huot L, Armoiry X, Gory B. EVIDENCE trial: design of a phase 2, randomized, controlled, multicenter study comparing flow diversion and traditional endovascular strategy in unruptured saccular wide-necked intracranial aneurysms. Neuroradiology. 2015 Jan;57(1):49-54. doi: 10.1007/s00234-014-1439-7. Epub 2014 Oct 4. PMID 25280445